CLINICAL TRIAL: NCT07193303
Title: The Immediate Effect of Mental Imagery on Upper Extremity Skills With the Patients of Parkinson's Disease
Brief Title: Mental Imagery on Upper Extremity Skills
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, Associate Profesor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: mental imagination
Record Dates: First submitted 2025-09-12; First posted 2025-09-25 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: PARKINSON DISEASE (Disorder); Mental Imagery; Motor Imagery
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1/study group (Experimental): Upper extremity skill tests will be performed on individuals diagnosed with idiopathic Parkinson's disease and recorded with a mental stopwatch using mental imagery.
  Interventions: Other: mental imagination
- 2/control group (No Intervention): Upper extremity skill tests will be performed on individuals diagnosed with idiopathic Parkinson's disease.

INTERVENTIONS:
Other: mental imagination — The Nine-Hole Peg Test (9 DPT) will be performed with a mental chronometer.the duration between actually physically performing the movement and mentally imagining the same movement will be recorded.
  Arms: 1/study group

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative disease, characterized pathologically by the progressive loss of dopaminergic neurons in the substantia nigra and clinically by the presence of motor symptoms such as bradykinesia, resting tremor, and/or rigidity. Among the motor deficits frequently observed in PD, patients are known to frequently report difficulties with manual dexterity. Many upper extremity and manual dexterity deficits are present in PD. Motor imagery (MI) is the imaginal execution of motor activities or the activation of specific muscles in the absence of any explicit feedback. This area of rehabilitation has been shown to be effective in improving and developing motor skills in many neurological conditions where patients exhibit motor recognition and execution impairments. MI can be applied at all stages of recovery from PD, is highly effective in movement-related pathologies, and can be performed independently.There is sufficient evidence that MI improves motor performance and learning in individuals with neurological disorders such as multiple sclerosis, stroke, and spinal cord injury. The study was designed to investigate the immediate effects of mental imagery, which is thought to be effective in controlling difficulties in planning and initiating movements in PD, on upper extremity skills. Therefore, the aim of this study was to determine the effect of mental imagery on upper extremity skills in PD.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged 40-75 years, diagnosed with idiopathic PD according to the UK Parkinson's Disease Association Brain Bank criteria by a specialist neurologist, with a Modified Hoehn & Yahr (m-HY) scale stage ≤4, and with a Mini Mental State Examination score of ≥24 for those with training and ≥18 for those without training, and with no known disease, volunteered to participate in the study.
* PD individuals with no other known neurological and/or systemic disease
* PD individuals without any upper extremity contractures

Exclusion Criteria:

* Individuals with diagnosed and/or treated psychiatric illnesses who are considered unable to complete the tests.
* Individuals who is taking neuroleptic medications or antidepressants.
* Individuals with orthopedic conditions that interfere with manual dexterity tests, such as severe dyskinesia, carpal tunnel syndrome, tendon injuries, or finger amputations; rheumatological conditions such as rheumatoid arthritis and osteoarthritis; and individuals with any neurological condition other than PD.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
The Nine-Hole Peg Test (9PPT) with Mental Chronometry | first day of the assesment
  Mental Chronometry: Mental chronometry is a method that measures imagery time, considered more objective than questionnaires in the assessment of MI. It examines the time difference between the actual physical execution of a movement and the mental image of the same movement.
  The Nine-Hole Peg Test (9PPT) is frequently used in the literature, although its validity and reliability as a mental chronometry test are lacking. In this task, the participant is required to remove nine pegs from the board to which they are fixed as quickly as possible and place them in a container on the board. The pegs used in the test (8 mm in diameter, 3 cm long) can be made of wood or plastic. The board (23 cm long, 10 cm wide, and 2 cm high) has a section at one end where the pegs are fixed (arranged in a 3x3 matrix) and a container-shaped space on the side for the pegs to be placed. Participants perform the test on both upper extremities. Before the test, all participants are given the opportunity to ho

SECONDARY OUTCOMES:
sosyodemographic form | first day of the assesment
  Medical history (disease duration and symptoms), demographic information, will be recorded.
Modified Hoehn & Yahr (m-HY) scale | first day of the assesment
  PD disability will be assessed with the m-HY scale. All of the patients with PD will be staged according to the Hoehn Yahr scale as follows: stage 1.0 (unilateral involvement only); stage 1.5 (unilateral and axial involvement); stage 2.0 (bilateral involvement without balance impairment); stage 2.5 (mild bilateral disease with improvement in the pull test); stage 3.0 (mild to moderate bilateral disease; some postural impairment; physically independent); stage 4.0 (severe disability; still able to walk or stand unaided).
Unified Parkinson's Disease Rating Scale (UPDRS) | first day of the asessment
  Symptom severity in PD is rated using the Unified Parkinson's Disease Rating Scale (UPDRS). Several items on this scale assess upper extremity and hand function. The Activities of Daily Living section assesses handwriting, cutting food, and grasping utensils. The Motor section assesses finger tapping, hand movements, and rapid alternating hand movements. These test items are scored from 0 to 4, with 4 representing maximum impairment and 0 representing normal movement ability. The UPDRS sections are subdivided into: Section I (mental dysfunction and mood); Section II (activities of daily living); Section III (motor); and Section IV (treatment-related complications).
Mini Mental State Examination (MMSE) | first day of the assessment
  This test was developed by Folstein in 1975. Its Turkish validity and reliability study was conducted by Güngen et al. in 2002. The MMSE, which is quite suitable for screening cognitive function in the elderly and assesses cognitive functions in five separate areas (orientation, registration, attention and calculation, recall, and language), is frequently used. A score below 24 on the MMSE indicates dementia, 24-26 indicates mild cognitive impairment, and 26 or above indicates normal cognitive function.
Muscle Strength Measurement | first day of the assesment
  Isometric strength will be measured using a digital muscle strength measurement device (KFORCE KINVENT) for the bilateral serratus anterior, upper trapezius, latissimus dorsi, deltoid, supraspinatus, teres minor, subscapularis, and biceps brachii muscles of the upper extremity.
Grip Strength Measurement | first day of the assesment
  A Jamar hand dynamometer (Baseline®) (and a PinchMeter (Baseline Mechanical Pinch Gauge with Case, Blue, 30 lb) will be used for grip strength measurement.
The Kinesthetic and Visual Imagery Questionnaire (KVIQ) | first day of the assesment
  The Kinesthetic and Visual Imagery Questionnaire (KVIQ), Short Form, was developed to determine the extent to which individuals visualize and feel imaged movements. It consists of a total of 10 movements measuring five visual and five kinesthetic imagery skills (23). The questionnaire is not a self-report measure but is administered by an assessor. All movements are assessed in a sitting position. The assessor first performs the relevant movement on themselves, and then the participant is asked to perform the same movement only once. The participant then imagines the movement and is asked to rate the visual clarity or intensity of sensations of the imagined movement using a five-point ordinal scale. Higher scores indicate greater visual clarity or intensity of sensations. This questionnaire will be used to assess mental imagery ability in our study.

CONTACTS AND LOCATIONS:
Overall Officials: hatice adıgüzel tat, Associate Professor, Study Chair — Kahramanmaras Sutcu Imam University; Asiya Uzun, Asisstant Prof, Principal Investigator — Kahramanmaras Sutcu Imam University; Yusuf Şinasi Kırmacı, Asisstant Prof, Study Chair — Kahramanmaras Sutcu Imam University; Abdulkadir Ertürk, Msc, Study Chair — Kahramanmaras Sutcu Imam University; Tuğçe Simay Özbay, Msc, Study Chair — Kahramanmaras Sutcu Imam University; Buket Tuğan Yıldız, Associate Professor, Study Chair — Kahramanmaras Sutcu Imam University; Deniz Tuncel, Proffessor, Study Chair — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaraş Sütçü imam University, Kahramanmaraş, Onikişubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No